CLINICAL TRIAL: NCT05691712
Title: A Randomized, Phase 3, Double Blind Trial Comparing the Effect of the Addition of Tirzepatide Versus the Addition of Placebo to Titrated Basal Insulin on Glycemic Control in Chinese Participants With Type 2 Diabetes
Brief Title: A Study of Tirzepatide (LY3298176) in Chinese Participants With Type 2 Diabetes
Acronym: SURPASS-CN-INS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18552; I8F-MC-GPIM (Other: Eli Lilly and Company)
Record Dates: First submitted 2023-01-11; First posted 2023-01-20 (Actual); Results first posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-07

CONDITIONS: Diabetes Type 2; Diabetes Mellitus; Glucose Metabolism Disorders; Metabolic Disease; Endocrine System Diseases
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Glucose Metabolism Disorders; Metabolic Diseases; Endocrine System Diseases | interventions — Tirzepatide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- 5 Milligram (mg) Tirzepatide (Experimental): Participants received 5 mg of tirzepatide administered as subcutaneous (SC) injection via a single-dose injection pen (SDP) once weekly (QW) for 40 weeks.
  The starting dose of tirzepatide was 2.5 mg QW, which increased by 2.5 mg every 4 weeks until the maintenance dose of 5 mg was reached.
  Interventions: Drug: Tirzepatide
- 10 mg Tirzepatide (Experimental): Participants received 10 mg of tirzepatide administered as SC injection via a SDP QW for 40 weeks.
  The starting dose of tirzepatide was 2.5 mg QW, which increased by 2.5 mg every 4 weeks (2.5 mg to 5 mg to 7.5 mg to 10 mg) until the maintenance dose of 10 mg was reached.
  Interventions: Drug: Tirzepatide
- 15 mg Tirzepatide (Experimental): Participants received 15 mg of tirzepatide administered as SC injection via a SDP QW for 40 weeks.
  The starting dose of tirzepatide was 2.5 mg QW, which increased by 2.5 mg every 4 weeks (2.5 mg to 5 mg to 7.5 mg to 10 mg to 12.5 mg to 15 mg) until the maintenance dose of 15 mg was reached.
  Interventions: Drug: Tirzepatide
- Placebo (Placebo Comparator): Participants received tirzepatide matched placebo administered as SC injection via a SDP QW for 40 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tirzepatide — Administered SC
  Other Names: LY3298176
  Arms: 10 mg Tirzepatide; 15 mg Tirzepatide; 5 Milligram (mg) Tirzepatide
Drug: Placebo — Administered SC
  Arms: Placebo

SUMMARY:
The main purpose of this study is to compare the effect of the addition of tirzepatide or placebo to titrated basal insulin on glycemic control in Chinese participants with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Have type 2 diabetes mellitus (T2DM)
* Have HbA1c ≥7.0% (53 mmol/mol) to ≤11% (97 mmol/mol)
* Have been treated with insulin glargine (U100) once daily alone, or in combination with metformin with or without SGLT-2i ≥90 days
* Have a body mass index (BMI) ≥23 kilograms per meter squared (kg/m²)

Exclusion Criteria:

* Have type 1 diabetes mellitus (T1DM)
* Have a history of chronic or acute pancreatitis
* Have proliferative diabetic retinopathy or diabetic macular edema or nonproliferative diabetic retinopathy that requires acute treatment
* Have a personal or family history of medullary thyroid carcinoma or personal history of multiple endocrine neoplasia syndrome type 2
* Have a history of severe hypoglycemia and/or hypoglycemia unawareness within the 6 months
* Have a history of diabetic ketoacidosis or hyperosmolar state/coma within the 6 months
* Have acute myocardial infarction, or cerebrovascular accident (stroke) or hospitalization due to congestive heart failure (CHF) in the past 2 months
* Have a serum calcitonin level of ≥35 ng/L, as determined by central laboratory
* Have acute or chronic hepatitis, signs, and symptoms of any other liver disease other than nonalcoholic fatty liver disease (NAFLD), or alanine aminotransferase (ALT) level >3.0 times the upper limit of normal (ULN), as determined by the central laboratory at study entry; participants with NAFLD are eligible for participation in this trial only if their ALT level is ≤3.0 times ULN.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 257 (Actual)
Dates: Start 2023-02-05 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (25):
- China (25):
  - The Second People's Hospital of Hefei, Hefei, Anhui
  - Beijing Hospital, Beijing, Beijing Municipality
  - Beijing Pinggu District Hospital, Beijing, Beijing Municipality
  - Chongqing General Hospital, Chongqing, Chongqing Municipality
  - Huizhou Municipal Central Hospital, Huizhou, Guangdong
  - The First Hospital of Harbin Medical University, Harbin, Heilongjiang
  - The Fourth Hospital of Harbin Medical University, Harbin, Heilongjiang
  - The First Affiliated Hospital of Henan University of Science &Technology, LuoyangShi, Henan
  - The Second Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - The First People's Hospital of Yueyang, Yueyang, Hunan
  - Baotou Central Hospital, Baotou, Inner Mongolia
  - Changzhou No.2 People's Hospital, Changzhou, Jiangsu
  - Nanjing First Hospital, Nanjing, Jiangsu
  - Zhongda Hospital Southeast University, Nanjing, Jiangsu
  - The Second Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - Wuxi People's Hospital, Wuxi, Jiangsu
  - The Affiliated Jiangyin Hospital of Southeast University Medical College, WuxiShi, Jiangsu
  - Affiliated Hospital of Jiangsu University, Zhenjiang, Jiangsu
  - The Third Hospital of Nanchang, Nanchang, Jiangxi
  - The First Affiliated Hospital of Xi'an Medical University, Xi'an, Shaanxi
  - Jinan Central Hospital, Jinan, Shandong
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Chengdu Fifth People's Hospital, Chengdu, Sichuan
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - Huzhou Central Hospital, Huzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: ata are available 6 months after the primary publication and approval of the indication studied in the US and European Union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Guo L, Dong X, Ma J, Liu M, Lu Y, Wang H, Li Q, Li L, Deng Y, Xu J. Efficacy and safety of tirzepatide added to basal insulin in patients with type 2 diabetes in China (SURPASS-CN-INS): a double-blind, multicentre, randomised, placebo-controlled, phase 3 trial. Lancet Diabetes Endocrinol. 2025 Dec;13(12):1015-1029. doi: 10.1016/S2213-8587(25)00248-7. Epub 2025 Oct 27. PMID 41167231

RESULTS

PARTICIPANT FLOW:
Groups:
- 5 Milligram (mg) Tirzepatide: Participants received 5 mg of tirzepatide administered as subcutaneous (SC) injection via a single-dose pen (SDP) once weekly (QW) for 40 weeks.
  The starting dose of tirzepatide was 2.5 mg QW, which increased by 2.5 mg every 4 weeks until the maintenance dose of 5 mg was reached.
Period: Overall Study
Arm/Group | 5 Milligram (mg) Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | Placebo
Started | 65 | 65 | 63 | 64
Received at Least One Dose of Study Drug | 65 | 65 | 63 | 64
Completed | 61 | 60 | 58 | 61
Not Completed | 4 | 5 | 5 | 3
Not completed — Adverse Event | 0 | 1 | 2 | 1
Not completed — Withdrawal by Subject | 2 | 3 | 3 | 1
Not completed — Death | 1 | 0 | 0 | 0
Not completed — Pregnancy | 0 | 1 | 0 | 0
Not completed — Assigned Treatment by Mistake | 1 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- 5 mg Tirzepatide: Participants received 5 mg of tirzepatide administered as SC injection via a SDP QW for 40 weeks.
  The starting dose of tirzepatide was 2.5 mg QW, which increased by 2.5 mg every 4 weeks until the maintenance dose of 5 mg was reached.
- Total: Total of all reporting groups
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | Placebo | Total
Number analyzed (Participants) | 65 | 65 | 63 | 64 | 257
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.10 (9.97) | 55.00 (11.58) | 55.80 (10.11) | 58.00 (10.24) | 56.70 (10.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 25 | 26 | 25 | 99
  Male | 42 | 40 | 37 | 39 | 158
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 65 | 65 | 63 | 64 | 257
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 65 | 65 | 63 | 64 | 257
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  China | 65 | 65 | 63 | 64 | 257
Percentage of Hemoglobin A1c (HbA1c) at Baseline [Mean (Standard Deviation); unit: Percentage of HbA1c] — HbA1c is the glycosylated fraction of hemoglobin A. HbA1c is measured primarily to identify average plasma glucose concentration over prolonged periods of time.
  Percentage of HbA1c | 8.64 (0.95) | 8.60 (1.09) | 8.75 (0.99) | 8.84 (0.99) | 8.71 (1.01)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in HbA1c (Tirzepatide 10 or 15 Milligram [mg])
Description: HbA1c is the glycosylated fraction of hemoglobin A. HbA1c is measured primarily to identify average plasma glucose concentration over prolonged periods of time. Least squares (LS) mean was calculated using mixed model repeated measures (MMRM) for post-baseline measures: Variable = Baseline + SGLT2i Use (Yes/No) + Treatment + Time + Treatment*Time (Type III sum of squares). Variance-Covariance structure (Actual Value) = Unstructured. Variance-Covariance structure (Change from Baseline) = Unstructured
Time Frame: Baseline, Week 40
Population: All randomized participants who received at least one dose of study drug with baseline and post-baseline value at the specified time point for this outcome excluding participants discontinuing study drug due to inadvertent enrollment and data after permanent discontinuation of study drug or initiation of rescue medication.
Measure: Least Squares Mean (Standard Error); unit: millimoles per mole (mmol/mol)
Arm/Group | 10 mg Tirzepatide | 15 mg Tirzepatide | Placebo
Number analyzed (Participants) | 57 | 55 | 58
millimoles per mole (mmol/mol) | -26.1 (1.367) | -25.9 (1.386) | -9.96 (1.340)
Statistical Analysis 1: Comparison: 10 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -16.1, 95% CI 2-sided [-19.9 to -12.36]
Statistical Analysis 2: Comparison: 15 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -15.9, 95% CI 2-sided [-19.7 to -12.10]

2. Secondary Outcome: Mean Change From Baseline in HbA1c (Tirzepatide 5 mg)
Description: HbA1c is the glycosylated fraction of hemoglobin A. HbA1c is measured primarily to identify average plasma glucose concentration over prolonged periods of time. LS mean was calculated using MMRM for post-baseline measures: Variable = Baseline + SGLT2i Use (Yes/No) + Treatment + Time + Treatment*Time (Type III sum of squares). Variance-Covariance structure (Actual Value) = Unstructured. Variance-Covariance structure (Change from Baseline) = Unstructured
Time Frame: Baseline, Week 40
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmol/mol
Arm/Group | 5 mg Tirzepatide | Placebo
Number analyzed (Participants) | 62 | 58
mmol/mol | -23.0 (1.329) | -9.96 (1.340)
Statistical Analysis 1: Comparison: 5 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -13.06, 95% CI 2-sided [-16.8 to -9.34]

3. Secondary Outcome: Mean Change From Baseline in Body Weight
Description: LSMean was calculated using MMRM for post-baseline measures: Variable = Baseline + Baseline HbA1c (<=8.0%, >8.0%) + SGLT2i Use (Yes/No) + Treatment + Time + Treatment*Time (Type III sum of squares). Variance-Covariance structure (Actual Value) = Unstructured. Variance-Covariance structure (Change from Baseline) = Unstructured
Time Frame: Baseline, Week 40
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: kilograms (kg)
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | Placebo
Number analyzed (Participants) | 62 | 57 | 55 | 58
kilograms (kg) | -2.7 (0.52) | -4.8 (0.54) | -4.3 (0.55) | 1.7 (0.53)
Statistical Analysis 1: Comparison: 5 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -4.4, 95% CI 2-sided [-5.8 to -2.9]
Statistical Analysis 2: Comparison: 10 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -6.5, 95% CI 2-sided [-8.0 to -5.0]
Statistical Analysis 3: Comparison: 15 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -6.0, 95% CI 2-sided [-7.5 to -4.5]

4. Secondary Outcome: Percentage of Participants With HbA1c <7.0% (53 Millimole/Mole [mmol/Mol]) and ≤6.5% (48 mmol/Mol)
Description: HbA1c is the glycosylated fraction of hemoglobin A. HbA1c is measured to identify average plasma glucose concentration over prolonged periods of time. The percentage of participants was calculated by dividing the number of participants reaching target HbA1c by the total number of participants analyzed, multiplied by 100. Percentage of Participants with HbA1c <7.0% (53 millimole/mole [mmol/mol]) and ≤6.5% (48 mmol/mol) is reported here.
Time Frame: Week 40
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | Placebo
Number analyzed (Participants) | 62 | 57 | 55 | 58
percentage of participants
  HbA1c <7.0% | 75.81 | 78.95 | 78.18 | 17.24
  HbA1c ≤6.5% | 59.68 | 77.19 | 69.09 | 6.90

5. Secondary Outcome: Mean Change From Baseline in Fasting Serum Glucose
Description: as for outcome 3
Time Frame: Baseline, Week 40
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: milligram per deciliter (mg/dL)
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | Placebo
Number analyzed (Participants) | 62 | 57 | 55 | 58
milligram per deciliter (mg/dL) | -45.5 (3.73) | -52.5 (3.87) | -51.0 (3.94) | -23.7 (3.84)
Statistical Analysis 1: Comparison: 5 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -21.9, 95% CI 2-sided [-32.4 to -11.3]
Statistical Analysis 2: Comparison: 10 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -28.9, 95% CI 2-sided [-39.6 to -18.1]
Statistical Analysis 3: Comparison: 15 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -27.3, 95% CI 2-sided [-38.2 to -16.5]

6. Secondary Outcome: Percentage of Participants With HbA1c <5.7% (39 mmol/Mol) [Tirzepatide 10 mg or 15 mg]
Description: HbA1c is the glycosylated fraction of hemoglobin A. HbA1c is measured to identify average plasma glucose concentration over prolonged periods of time. Percentage of participants with HbA1c <5.7% (39 mmol/Mol) is reported here.
Time Frame: Week 40
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | 10 mg Tirzepatide | 15 mg Tirzepatide | Placebo
Number analyzed (Participants) | 57 | 55 | 58
percentage of participants | 17.54 | 25.45 | 0.00

7. Secondary Outcome: Percentage of Participants With HbA1c <5.7% (39 mmol/Mol) [Tirzepatide 5 mg]
Description: as for outcome 6
Time Frame: Week 40
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | 5 mg Tirzepatide | Placebo
Number analyzed (Participants) | 62 | 58
percentage of participants | 9.68 | 0.00

8. Secondary Outcome: Mean Change From Baseline in Daily Average 7-point Self-monitored Blood Glucose Profiles
Description: The SMBG data were collected at the following 7 time points: Morning Premeal - Fasting, Morning 2-hour Post meal, Midday Premeal, Midday 2-hour Post meal, Evening Premeal, Evening 2-hour Post meal and Bedtime. The daily average was calculated as the average of the 7 blood glucose values collected on a particular day. LS Mean was calculated using MMRM for post-baseline measures: Variable = Baseline + Baseline HbA1c (<=8.0%, >8.0%) + SGLT2i Use (Yes/No) + Treatment + Time + Treatment*Time (Type III sum of squares). Variance-Covariance structure (Actual Value) = Unstructured. Variance-Covariance structure (Change from Baseline) = Unstructured.
Time Frame: Baseline, Week 40
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: millimoles per liter per day(mmol/L/day)
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | Placebo
Number analyzed (Participants) | 62 | 57 | 55 | 63
millimoles per liter per day(mmol/L/day)
  Morning Premeal - Fasting: number analyzed (Participants) | 61 | 56 | 53 | 57
  Morning Premeal - Fasting | -2.62 (0.127) | -2.53 (0.132) | -2.80 (0.136) | -2.22 (0.131)
  Morning 2-hour Postmeal: number analyzed (Participants) | 56 | 54 | 51 | 55
  Morning 2-hour Postmeal | -4.78 (0.300) | -5.34 (0.306) | -5.05 (0.313) | -2.57 (0.300)
  Midday Premeal: number analyzed (Participants) | 61 | 56 | 53 | 57
  Midday Premeal | -2.87 (0.247) | -3.52 (0.258) | -3.26 (0.263) | -1.32 (0.253)
  Midday 2-hour Postmeal: number analyzed (Participants) | 57 | 55 | 51 | 55
  Midday 2-hour Postmeal | -4.05 (0.318) | -4.10 (0.325) | -3.65 (0.335) | -1.46 (0.322)
  Evening Premeal | -2.84 (0.264) | -3.64 (0.276) | -3.20 (0.285) | -0.95 (0.271)
  Evening 2-hour Postmeal: number analyzed (Participants) | 55 | 55 | 49 | 54
  Evening 2-hour Postmeal | -3.97 (0.347) | -4.52 (0.351) | -4.42 (0.367) | -1.47 (0.346)
  Bedtime: number analyzed (Participants) | 60 | 56 | 52 | 54
  Bedtime | -3.41 (0.287) | -4.19 (0.297) | -3.85 (0.307) | -1.71 (0.298)

9. Secondary Outcome: Percentage of Participants Who Achieved Weight Loss of ≥5%
Description: Percentage of Participants who Achieved Weight Loss ≥5% is reported here.
Time Frame: Week 40
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | Placebo
Number analyzed (Participants) | 62 | 57 | 55 | 58
percentage of participants | 25.81 | 49.12 | 60.00 | 1.72

10. Secondary Outcome: Percentage of Participants Who Achieved Weight Loss of ≥10%
Description: Percentage of Participants who Achieved Weight Loss ≥10% is reported here.
Time Frame: Week 40
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | Placebo
Number analyzed (Participants) | 62 | 57 | 55 | 58
percentage of participants | 8.06 | 21.05 | 25.45 | 0.00

11. Secondary Outcome: Percentage of Participants Who Achieved Weight Loss of ≥15%
Description: Percentage of Participants who Achieved Weight Loss ≥15% is reported here.
Time Frame: Week 40
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | Placebo
Number analyzed (Participants) | 62 | 57 | 55 | 58
percentage of participants | 4.84 | 5.26 | 9.09 | 0.00

12. Secondary Outcome: Percent Change From Baseline in Daily Mean Insulin Glargine Dose
Description: LS Mean was calculated using MMRM for post-baseline measures: log(Actual Measurement/Baseline) = log(Baseline) + Baseline HbA1c (<=8.0%, >8.0%) + SGLT2i Use (Yes/No) + Treatment + Time + Treatment*Time (Type III sum of squares). Variance-Covariance structure (Change from Baseline) = Unstructured.
Time Frame: Baseline, Week 40
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | Placebo
Number analyzed (Participants) | 62 | 57 | 55 | 58
percent change | 23.90 (6.424) | 21.95 (6.471) | 18.21 (6.364) | 69.28 (8.826)

13. Secondary Outcome: Percentage of Participants With HbA1c <7.0%, Without Weight Gain (<0.1 Kilogram [kg]) and Without Hypoglycemia, (Blood Glucose <3.0 mmol/L <54 Milligram/Deciliter [mg/dL])
Description: Percentage of Participants with HbA1c <7.0%, Without Weight Gain (<0.1 Kilogram [kg]) and Without Hypoglycemia, (Blood Glucose <3.0 mmol/L <54 Milligram/Deciliter [mg/dL]) is reported here
Time Frame: Week 40
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | Placebo
Number analyzed (Participants) | 62 | 57 | 55 | 58
percentage of participants | 59.68 | 70.18 | 67.27 | 5.17

14. Secondary Outcome: Percentage of Participants With HbA1c ≤6.5%, Without Weight Gain <0.1 kg and Without Hypoglycemia (Blood Glucose <3.0 mmol/L [54 mg/dL])
Description: Percentage of Participants with HbA1c ≤6.5%, Without Weight Gain <0.1 kg and Without Hypoglycemia (Blood glucose <3.0 mmol/L [54 mg/dL]) is reported here.
Time Frame: Week 40
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | Placebo
Number analyzed (Participants) | 62 | 57 | 55 | 58
percentage of participants | 46.77 | 70.18 | 61.82 | 1.72

15. Secondary Outcome: Percentage of Participants With HbA1c <7.0%, Without Weight Gain <0.1 kg and Without Hypoglycemia (Blood Glucose <3.9 mmol/L [70 mg/dL] or Severe Hypoglycemia)
Description: Percentage of Participants with HbA1c <7.0%, Without Weight Gain <0.1 kg and Without Hypoglycemia (Blood Glucose <3.9 mmol/L [70 mg/dL] or Severe Hypoglycemia) is reported here.
Time Frame: Week 40
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | Placebo
Number analyzed (Participants) | 62 | 57 | 55 | 58
percentage of participants | 51.61 | 57.89 | 47.27 | 5.17

16. Secondary Outcome: Percentage of Participants With HbA1c ≤6.5%, Without Weight Gain <0.1 kg and Without Hypoglycemia (Blood Glucose <3.9 mmol/L [70 mg/dL] or Severe Hypoglycemia)
Description: Percentage of Participants with HbA1c ≤6.5%, Without Weight Gain <0.1 kg and Without Hypoglycemia (Blood glucose <3.9 mmol/L [70 mg/dL] or Severe Hypoglycemia) is reported here.
Time Frame: Week 40
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | Placebo
Number analyzed (Participants) | 62 | 57 | 55 | 58
percentage of participants | 38.71 | 57.89 | 43.64 | 1.72

ADVERSE EVENTS:
Time Frame: Baseline up to week 44
Description: All randomized participants who received at least one dose of study drug regardless of adherence to study drug or initiation of rescue medication. Based on the planned safety analysis, adverse events were collected per the treatment regimen, irrespective of each dose level. Gender specific events only occurring in male or female participants have had the number of participants At Risk adjusted accordingly.
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | Placebo
All-Cause Mortality (participants affected / at risk) | 1/65 | 0/65 | 0/63 | 0/64
Serious Adverse Events (participants affected / at risk) | 8/65 | 5/65 | 8/63 | 7/64
Other Adverse Events (participants affected / at risk) | 45/65 | 49/65 | 49/63 | 31/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | 5 mg Tirzepatide (N=65) | 10 mg Tirzepatide (N=65) | 15 mg Tirzepatide (N=63) | Placebo (N=64)
Arteriosclerosis coronary artery (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Deafness neurosensory (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 1 (2) | 0 (0) | 1 (2) | 1 (1)
Diabetic retinopathy (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epiretinal membrane (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye disorder (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Retinal detachment (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vitreous haemorrhage (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chronic gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mass (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sudden death (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Soft tissue infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Synovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colorectal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ovarian cyst (Reproductive system and breast disorders) | 0/23 (0) | 0/25 (0) | 1/26 (1) | 0/25 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | 5 mg Tirzepatide (N=65) | 10 mg Tirzepatide (N=65) | 15 mg Tirzepatide (N=63) | Placebo (N=64)
Palpitations (Cardiac disorders) | 0 (0) | 4 (4) | 0 (0) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 7 (7) | 3 (3) | 4 (5) | 0 (0)
Constipation (Gastrointestinal disorders) | 4 (4) | 2 (2) | 2 (2) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 17 (61) | 24 (45) | 23 (44) | 5 (10)
Dyspepsia (Gastrointestinal disorders) | 4 (7) | 0 (0) | 2 (2) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3) | 7 (8) | 7 (13) | 2 (2)
Toothache (Gastrointestinal disorders) | 3 (3) | 2 (2) | 0 (0) | 4 (5)
Vomiting (Gastrointestinal disorders) | 4 (7) | 6 (7) | 4 (20) | 0 (0)
Fatigue (General disorders) | 0 (0) | 4 (4) | 1 (1) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 13 (17) | 11 (14) | 11 (12) | 9 (11)
Amylase increased (Investigations) | 4 (6) | 8 (11) | 3 (3) | 2 (3)
Blood creatine phosphokinase increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 4 (4)
Lipase increased (Investigations) | 12 (15) | 14 (19) | 6 (6) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 19 (23) | 16 (22) | 20 (33) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 2 (2) | 5 (5) | 3 (3) | 4 (4)
Hyperuricaemia (Metabolism and nutrition disorders) | 4 (4) | 3 (4) | 6 (6) | 2 (2)
Headache (Nervous system disorders) | 3 (3) | 4 (4) | 0 (0) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 2/42 (2) | 2/40 (2) | 0/37 (0) | 0/39 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2023-11-17): https://cdn.clinicaltrials.gov/large-docs/12/NCT05691712/Prot_000.pdf
  • Statistical Analysis Plan (2025-01-08): https://cdn.clinicaltrials.gov/large-docs/12/NCT05691712/SAP_001.pdf